CLINICAL TRIAL: NCT02458924
Title: Niacin Skin Flush Response in Patients With Schizophrenia, Their First Degree Relatives, Bipolar Disorder Patients, and Healthy Controls
Brief Title: Niacin Skin Flush Response in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Maryam Tabatabaeian, Dr., Isfahan University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 393230
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — methyl nicotinate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Schizophrenia (Active Comparator): Skin niacin test was performed by two concentrations including 0.5 ml solutions of 0.01 M and 0.1 M diluted methyl nicotinate. The two solutions were applied for one minute to the inside of the different forearms of each individual.
  Interventions: Biological: Niacin skin test
- Bipolar disorder (Active Comparator): Skin niacin test was performed by two concentrations including 0.5 ml solutions of 0.01 M and 0.1 M diluted methyl nicotinate. The two solutions were applied for one minute to the inside of the different forearms of each individual.
  Interventions: Biological: Niacin skin test
- First degree relatives (Active Comparator): Skin niacin test was performed by two concentrations including 0.5 ml solutions of 0.01 M and 0.1 M diluted methyl nicotinate. The two solutions were applied for one minute to the inside of the different forearms of each individual.
  Interventions: Biological: Niacin skin test
- Health controls (Active Comparator): Skin niacin test was performed by two concentrations including 0.5 ml solutions of 0.01 M and 0.1 M diluted methyl nicotinate. The two solutions were applied for one minute to the inside of the different forearms of each individual.
  Interventions: Biological: Niacin skin test

INTERVENTIONS:
Biological: Niacin skin test — Two concentrations including 0.5 ml solutions of 0.01 M and 0.1 M diluted methyl nicotinate were applied for one minute to the inside of the different forearms of each individual.
  Other Names: Methyl nicotinate

SUMMARY:
Patients with schizophrenia have abnormal skin flush response to niacin, but the niacin skin test accuracy is not well studied in these patients. The study evaluated the niacin skin test accuracy in adult hospitalized schizophrenia patients and their first degree relatives, bipolar disorder patients, and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia patients and bipolar disorder patients diagnosed according to the Diagnostic and Statistical Manual of Mental Disorders version IV criteria
* Normal healthy subjects without a psychiatric history
* First degree relatives of schizophrenic patients

Exclusion Criteria:

* Dermatological lesions, asthma or allergic disease, diabetes, chronic hypertension, vasculitis, substance use disorders (except cigarette smoking), or pregnancy
* Taking any oral medication that could affect the metabolism of prostaglandins such as nonsteroidal anti-inflammatory drugs or corticosteroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Skin flush response | Every 5 minutes for 20 minutes
  Skin response was assessed by a single physician every 5 minutes for 20 minutes after removal of the substance. The outcome assessor was not blinded to the applied solution dosages. The strength of the flushing reaction was classified as 0 = no redness, 1 = faint redness, 2 = distinct redness, and 3 = extreme or maximum redness.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Tabatabaeian, MD, Principal Investigator — Isfahan University of Medical Sciences